CLINICAL TRIAL: NCT02372383
Title: Pharmacokinetic Evaluation of Nontuberculous Mycobacterial Antibiotics in Cystic Fibrosis Versus Controls
Brief Title: Improving Treatment of Nontuberculous Mycobacterial Infection in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-1043; UL1TR001082 (NIH)
Record Dates: First submitted 2014-06-20; First posted 2015-02-26 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pharmacokinetics; Pharmacodynamics; Nontuberculous Mycobacteria; Treatment
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ethambutol; Rifampin; Azithromycin; Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fasting (Experimental): Subjects with CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes
  * Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg)
  * Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg)
  * Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg)
  Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Interventions: Drug: Ethambutol; Drug: Rifampin; Drug: Azithromycin
- Food/Enzymes (Experimental): Subjects with CF will be given the antimycobacterial drugs with a standardized meal plus a typical meal-dose of pancreatic enzymes (Pancrelipase).
  * Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg)
  * Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg)
  * Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg)
  Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Interventions: Drug: Ethambutol; Drug: Rifampin; Drug: Azithromycin; Drug: Pancrelipase
- Healthy Controls (Active Comparator): Healthy subjects without CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes
  * Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg)
  * Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg)
  * Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg)
  Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Interventions: Drug: Ethambutol; Drug: Rifampin; Drug: Azithromycin

INTERVENTIONS:
Drug: Ethambutol — Anti-mycobacterial oral drug
  Other Names: Myambutol
Drug: Rifampin — Anti-mycobacterial oral drug
  Other Names: Rifadin
Drug: Azithromycin — Anti-mycobacterial oral drug
  Other Names: Zithromax
Drug: Pancrelipase — Pancreatic enzyme replacement therapy
  Other Names: Creon; Zenpep; Pertzye
  Arms: Food/Enzymes

SUMMARY:
The purpose of this study is to determine antimycobacterial drug pharmacokinetics (PK) and pharmacodynamics (PD) in patients with cystic fibrosis (CF) to improve treatment of nontuberculous mycobacterial (NTM) lung disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine antimycobacterial drug pharmacokinetics (PK) and pharmacodynamics (PD) in patients with cystic fibrosis (CF) to improve treatment of nontuberculous mycobacterial (NTM) lung disease.

Aim 1: Determine the PK profile of oral antimycobacterial drugs (azithromycin, rifampin and ethambutol) under both fasting conditions and when taken with food plus supplemental pancreatic enzymes in subjects with pancreatic insufficient, compared to healthy controls.

Aim 2: Begin to investigate the influence of inflammation, host characteristics, and drug metabolism on the PK of the antimycobacterial drugs.

Aim 3: Estimate an optimized dosing regimen for the antimycobacterial drugs against Mycobacterium avium complex (MAC) using historic minimum inhibitory concentration (MIC) data and models of Mycobacterium tuberculosis or MAC infection.

The central goal of this study is to improve treatment of NTM infection in CF. Upon completion of this study the investigators will determine if and why PK of the antimycobacterial drugs are altered in CF. More importantly, the investigators will develop CF-specific guidelines to achieve therapeutic goals with recommendations for drug dosing (including dose, dose frequency and timing in relation to meals and supplemental pancreatic enzymes) and timing of therapeutic monitoring to be used for future treatment of NTM lung disease in CF.

ELIGIBILITY:
CF Subject Inclusion Criteria:

* CF diagnosis defined as a sweat chloride >60mEq/L and/or the presence of two disease-causing CFTR mutations.
* Ages 16 years and above.
* Pancreatic insufficient status defined as previous fecal pancreatic elastase <100mcg/g stool and/or having 2 disease-causing CFTR mutations known to be associated with pancreatic insufficiency, and taking supplemental pancreatic enzymes between 1000-2500 lipase units/kg/meal.
* No positive NTM cultures in the last 2 years.
* Pulmonary function: Most recent FEV1 > 40% predicted.
* Willing to participate in and comply with the study procedures, and willingness of a parent or legally authorized representative to provide written informed consent for those subjects less than 18 years of age.

Healthy Control Inclusion Criteria:

* Ages 18 years and above.
* BMI below 30 to best match CF body type.
* Willing to participate in and comply with the study procedures, and willingness of a parent or legally authorized representative to provide written informed consent for those subjects less than 18 years of age.

CF Subject Exclusion Criteria:

* Allergy or intolerance to rifampin, ethambutol, or azithromycin.
* Hepatic insufficiency defined as having an AST or ALT greater than three times the upper limit of normal at the screening appointment.
* Previous surgical bowel resection.
* Previous lung transplant.
* Use of medications known to interact with the antimycobacterial drug levels; of note, the most common interactions in CF patients are the use of itraconazole, voriconazole, and ivacaftor. We will have subjects hold H2 blockers and proton pump inhibitors for 3 days prior to each PK study day.
* Inability to hold azithromycin: Subjects will not be excluded if they are on chronic azithromycin for immunomodulatory purposes; however, we will ask that the subjects hold the azithromycin starting at the screening visit, through a 2 week wash-out period prior to Visit 2, and remain off through the end of Visit 3 (about 4 weeks total).
* Acute exacerbations: exclusion if any addition of oral, IV, or inhaled antibiotics, or an acute gastrointestinal illness with vomiting or diarrhea in the 2 weeks prior to each visit. No exclusion for previously prescribed alternating chronic inhaled or oral antibiotics.
* We will also exclude pregnant women (urine pregnancy test will be performed for females on the day of each PK study) and decisionally challenged subjects.

Healthy Control Exclusion Criteria:

* Allergy or intolerance to rifampin, ethambutol, or azithromycin.
* Hepatic insufficiency defined as having an AST or ALT greater than three times the upper limit of normal at the screening appointment.
* Previous chronic GI disease or surgical bowel resection.
* Use of medications known to interact with the antimycobacterial drug levels. We will have subjects hold H2 blockers and proton pump inhibitors for 3 days prior to the PK study day.
* Acute illness: exclusion if respiratory illness requiring antibiotics or gastrointestinal illness with vomiting or diarrhea in the 2 weeks prior to the PK visit.
* We will also exclude pregnant women (urine pregnancy test will be performed on the day of PK study) and decisionally challenged subjects.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Martiniano, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colroado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martiniano SL, Wagner BD, Brennan L, Wempe MF, Anderson PL, Daley CL, Anthony M, Nick JA, Sagel SD. Pharmacokinetics of oral antimycobacterials and dosing guidance for Mycobacterium avium complex treatment in cystic fibrosis. J Cyst Fibros. 2021 Sep;20(5):772-778. doi: 10.1016/j.jcf.2021.04.011. Epub 2021 May 21. PMID 34030986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 CF subjects and 10 Healthy controls will be studied
Groups:
- Healthy Controls (Fasting Only): Healthy subjects without CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes
  * Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg)
  * Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg)
  * Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg)
  Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Ethambutol: Anti-mycobacterial oral drug
  Rifampin: Anti-mycobacterial oral drug
  Azithromycin: Anti-mycobacterial oral drug
- CF Patients, Fasting, Then Food: Fasting for 1 day, then washout for 2 weeks, then Food for 1 day.
  Subjects with CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg) Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg) Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg) Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Experimental: Food/Enzymes Subjects with CF will be given the antimycobacterial drugs with a standardized meal plus a typical meal-dose of pancreatic enzymes (Pancrelipase).
  Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg) Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg) Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg) Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
- CF Patients, Food Then Fasting: Food for 1 day, then washout for 2 weeks, then Fasting for 1 day.
  Subjects with CF will be given the antimycobacterial drugs with a standardized meal plus a typical meal-dose of pancreatic enzymes (Pancrelipase).
  Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg) Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg) Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg) Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Subjects with CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg) Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg) Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg) Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
Period: First Intervention (1 Day)
Arm/Group | Healthy Controls (Fasting Only) | CF Patients, Fasting, Then Food | CF Patients, Food Then Fasting
Started | 10 | 11 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 1 | 0
Not completed — Unable to collect blood | 0 | 1 | 0
Period: Washout (14 Days)
Arm/Group | Healthy Controls (Fasting Only) | CF Patients, Fasting, Then Food | CF Patients, Food Then Fasting
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Healthy Controls (Fasting Only) | CF Patients, Fasting, Then Food | CF Patients, Food Then Fasting
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One patient was unable to participate at day 1 from the CF Subjects arm, and baseline data was not collected. Baseline demographics data was not stratified between the "Fasting, then Food" versus "Food, then Fasting" sequences. Baseline data was only collected for Healthy Controls versus CF subjects.
Groups:
- CF Subjects: Fasting State Subjects with CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes
  * Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg)
  * Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg)
  * Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg)
  Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Ethambutol: Anti-mycobacterial oral drug
  Rifampin: Anti-mycobacterial oral drug
  Azithromycin: Anti-mycobacterial oral drug
  Food/Enzymes State Subjects with CF will then cross-over and be given the same dose of the 3 antimycobacterial drugs with a standardized meal plus a typical meal-dose of pancreatic enzymes (Pancrelipase). CF subjects will be randomized to either receive the medications in the Fasting or Food/Enzymes state first.
- Total: Total of all reporting groups
Arm/Group | CF Subjects | Healthy Controls (Fasting Only) | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 19 | 10 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 18.3 [16.1 to 24.8] | 25.3 [18.2 to 30.7] | 20.6 [16.1 to 30.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 13 | 4 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Median Maximal Drug Concentration (Cmax)
Description: Cmax of the oral antimycobacterial drugs (azithromycin, rifampin and ethambutol) under both fasting conditions and when taken with food plus supplemental pancreatic enzymes in subjects with pancreatic insufficient CF, compared to healthy controls.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
Measure: Median (Full Range); unit: mg/L
Groups:
- Healthy Controls: Healthy subjects without CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes
  * Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg)
  * Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg)
  * Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg)
  Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Ethambutol: Anti-mycobacterial oral drug
  Rifampin: Anti-mycobacterial oral drug
  Azithromycin: Anti-mycobacterial oral drug
- CF Fasting; CF Food: Subjects with CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes
  * Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg)
  * Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg)
  * Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg)
  Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Ethambutol: Anti-mycobacterial oral drug
  Rifampin: Anti-mycobacterial oral drug
  Azithromycin: Anti-mycobacterial oral drug
  CF subjects will then cross-over following at least a 2 week washout time point and and be given the same dose of the 3 antimycobacterial drugs with a standardized meal plus a typical meal-dose of pancreatic enzymes (Pancrelipase).
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 20
mg/L
  Rifampin | 16.56 [10.2 to 27.0] | 12.5 [6.6 to 21.9] | 11.2 [4.7 to 14.5]
  Ethambutol | 3.0 [2.3 to 4.7] | 4.2 [1.1 to 6.8] | 4.3 [1.0 to 5.7]
  Azithromycin | 1.1 [0.6 to 2.1] | 2.0 [0.1 to 5.3] | 2.2 [0.1 to 4.1]

2. Secondary Outcome: Other PK Measures: Median Time to Maximal Drug Concentration (Tmax)
Description: Tmax of the oral antimycobacterial drugs (azithromycin, rifampin and ethambutol) under both fasting conditions and when taken with food plus supplemental pancreatic enzymes in subjects with pancreatic insufficient CF, compared to healthy controls
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
Measure: Median (Full Range); unit: hours
Groups:
- CF Patients, Fasting; CF Patients, Food: Subjects with CF will be given the antimycobacterial drugs in the fasting state, without supplemental pancreatic enzymes
  * Rifampin 10mg/kg oral once daily (max 600mg, round to closest 150mg)
  * Ethambutol 15mg/kg oral once daily (max 2500mg, round to nearest 100mg)
  * Azithromycin 10mg/kg oral once daily (max 500mg, rounded to the nearest 250mg)
  Blood will be drawn at time points 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
  Ethambutol: Anti-mycobacterial oral drug
  Rifampin: Anti-mycobacterial oral drug
  Azithromycin: Anti-mycobacterial oral drug
  CF subjects will then cross-over following at least a 2 week washout time point and and be given the same dose of the 3 antimycobacterial drugs with a standardized meal plus a typical meal-dose of pancreatic enzymes (Pancrelipase).
Arm/Group | Healthy Controls | CF Patients, Fasting | CF Patients, Food
Number analyzed (Participants) | 10 | 20 | 20
hours
  Rifampin | 1.5 [1 to 4] | 1.5 [1 to 3] | 2.5 [1 to 6]
  Ethambutol | 2.3 [1 to 4] | 2.3 [1 to 4] | 2.0 [1 to 4]
  Azithromycin | 2.0 [1 to 3] | 2.0 [1 to 4] | 2.0 [1 to 4]

3. Secondary Outcome: Other PK Measures: Half-life (t1/2)
Description: t1/2 of the oral antimycobacterial drugs (azithromycin, rifampin and ethambutol) under both fasting conditions and when taken with food plus supplemental pancreatic enzymes in subjects with pancreatic insufficient CF, compared to healthy controls
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
Measure: Median (Full Range); unit: hours
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 20
hours
  Rifampin | 3.8 [2.6 to 7.0] | 3.4 [2.2 to 5.9] | 3.4 [2.3 to 8.0]
  Ethambutol | 5.3 [3.3 to 6.0] | 4.3 [3.1 to 7.2] | 4.7 [3.0 to 15.1]
  Azithromycin | 6.2 [3.3 to 7.0] | 5.2 [2.5 to 14.0] | 6.6 [2.5 to 14.4]

4. Secondary Outcome: Other PK Measures: Drug Clearance
Description: drug clearance of the oral antimycobacterial drugs (azithromycin, rifampin and ethambutol) under both fasting conditions and when taken with food plus supplemental pancreatic enzymes in subjects with pancreatic insufficient CF, compared to healthy controls
  Reported here are the Median (range) CL in the CF fasting state compared to HC for Rifampin.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
Measure: Median (Full Range); unit: L/h
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 20
L/h
  Rifampin | 5.1 [3.8 to 8.5] | 7.9 [3.6 to 15.7] | 7.6 [4.4 to 19.5]
  Ethambutol | 45.3 [34.3 to 61.8] | 42.4 [23.6 to 156.6] | 37.3 [27.7 to 185.2]
  Azithromycin | 88.6 [40.3 to 190.9] | 73.6 [31.9 to 978.8] | 82.8 [41.7 to 567.5]

5. Secondary Outcome: Other PK Measures: Volume of Distribution (Vd)
Description: Vd of the oral antimycobacterial drugs (azithromycin, rifampin and ethambutol) under both fasting conditions and when taken with food plus supplemental pancreatic enzymes in subjects with pancreatic insufficient CF, compared to healthy controls
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
Measure: Median (Full Range); unit: L
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 20
L
  Rifampin | 31.3 [16.4 to 39.0] | 39.7 [21.3 to 67.5] | 37.4 [25.9 to 105.6]
  Ethambutol | 352.8 [162.0 to 453.0] | 274.6 [139.7 to 1045.9] | 354.3 [147.3 to 1866.4]
  Azithromycin | 717.0 [406.1 to 1083.4] | 549.2 [201.5 to 9503.5] | 621.3 [249.3 to 8608.7]

6. Secondary Outcome: Covariates of PK Measures: C-reactive Protein (CRP)
Description: Median Concentration of C-reactive Protein. Begin to investigate the influence of inflammation, host characteristics, and drug metabolism on the PK of the antimycobacterial drugs.
Time Frame: baseline
Population: This Outcome Measure was only analyzed at the Fasting period and was not collected during the Food period of the study. Therefore, 0 participants are analyzed for the "CF Food" arm for this Outcome Measure.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 0
mg/dL | 0.2 [0.0 to 5.1] | 0.8 [0.2 to 9] |

7. Secondary Outcome: Covariates of PK Measures: Circulating Neutrophil Count
Description: Circulating neutrophil count. Begin to investigate the influence of inflammation, host characteristics, and drug metabolism on the PK of the antimycobacterial drugs
Time Frame: baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: 10^3 cells/uL
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 0
10^3 cells/uL | 3.0 [1.4 to 7.2] | 3.8 [2.5 to 7.7] |

8. Secondary Outcome: Covariates of PK Measures: Body Mass Index
Description: Body mass index (BMI). Begin to investigate the influence of inflammation, host characteristics, and drug metabolism on the PK of the antimycobacterial drugs
Time Frame: baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: kg/m^2
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 0
kg/m^2 | 23.0 [18.9 to 25.1] | 21.9 [18.0 to 26.6] |

9. Secondary Outcome: Covariates of PK Measures: Creatinine
Description: Creatinine. Begin to investigate the influence of inflammation, host characteristics, and drug metabolism on the PK of the antimycobacterial drugs
Time Frame: baseline
Population: as for outcome 6
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 0
mg/dL | 1.0 [0.8 to 1.2] | 0.9 [0.7 to 1.1] |

10. Secondary Outcome: Area Under the Curve (AUC)
Description: AUC of the oral antimycobacterial drugs (azithromycin, rifampin and ethambutol) under both fasting conditions and when taken with food plus supplemental pancreatic enzymes in subjects with pancreatic insufficient CF, compared to healthy controls.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post dose
Measure: Median (Full Range); unit: mg*h/L
Arm/Group | Healthy Controls | CF Fasting | CF Food
Number analyzed (Participants) | 10 | 20 | 20
mg*h/L
  Rifampin | 118.3 [70.5 to 156] | 76 [38.1 to 167.5] | 79.2 [30.8 to 136.7]
  Ethambutol | 21.4 [16.2 to 30.4] | 21.8 [6.4 to 38.2] | 23.6 [5 to 36]
  Azithromycin | 5.6 [2.6 to 12.4] | 6.8 [0.5 to 15.7] | 6 [0.9 to 12]

ADVERSE EVENTS:
Time Frame: During the time of participation in the study, about 6 weeks.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. One participant is included in the Fasting arm who dropped out immediately after, prior to the Food period.
Arm/Group | Healthy Controls | CF Patients, Fasting | CF Patients, Food
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes